CLINICAL TRIAL: NCT04247685
Title: Evaluation of MRI-conditional 12-lead ECG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Graham Wright (Other)
Responsible Party: Sponsor-Investigator, Dr. Graham Wright, Senior scientist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 314-2019
Record Dates: First submitted 2019-10-28; First posted 2020-01-30 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The investigators will aim to recruit 2-3 patients per month, with a total of 40 patients over two years. These 40 patients will be assigned into two MRI groups -12-lead ECG gating system as the study group and 3-lead ECG gating system as the control group. The study group patients will have MRI with 12-lead ECG monitoring device produced by a Massachusetts-based medical device company MiRTLE Medical, while the control group will have MRI with 3-lead ECG gating which is standard of care. Diagnostic image quality and severity of artifact will be evaluated to compare these two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-Lead ECG (Experimental): The study group patients will have MRI with 12-lead ECG monitoring device produced by a Massachusetts-based medical device company MiRTLE Medical
  Interventions: Device: 12-lead ECG monitoring device (MiRTLE Medical)
- 3-lead ECG gating system (Active Comparator): the control group will have MRI with 3-lead ECG gating which is standard of care.
  Interventions: Device: 3-lead ECG gating system

INTERVENTIONS:
Device: 12-lead ECG monitoring device (MiRTLE Medical) — 12-lead ECG monitoring device produced by a Massachusetts-based medical device company MiRTLE Medical is the experimental device;
  Arms: 12-Lead ECG
Device: 3-lead ECG gating system — 3-lead ECG gating system is the placebo/standard of care
  Arms: 3-lead ECG gating system

SUMMARY:
With MRI's increasing role in detecting central nervous system and orthopedic diseases, patients with ischemic history are increasingly referred for MRI exams. Currently, 3-lead ECG gating systems are utilized during cardiac MRI scanning as standard of care. However, this monitoring system is often insufficient to evaluate for the development of important arrhythmias or ischemia during MRI scanning. Morevoer, MRI associated magnetic fields and radio frequency pulses can produce interference in the ECG signal that leads to non-diagnostic ECG signals. MiRTLE Medical, a Massachusetts-based medical device company, has developed a high-fidelity, MRI-conditional 12-lead ECG monitoring system. This 12-lead ECG system is a first of its kind that addresses the MRI-induced interference and safety issues. This study is to evaluate the efficacy of this 12-lead ECG system in the clinical setting. The investigators hope that this system will be helpful for image-guided therapeutics especially electrophysiology.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Atrial fibrillation
* Provision of informed consent
* Eligible for the Ontario Health Insurance Plan

Exclusion Criteria:

* Failure to provide informed consent
* Pregnant women
* CMR contra-indicated
* Hemodynamically unstable
* Permanent pacemaker/ICD
* Aneurysm clip/carotid artery vascular clamp
* Claustrophobic

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
absolute numbers and percentages | up to 6 weeks
  the following patient data will be collected as absolute numbers and percentages in a future Table 1: Age, Sex, Cardiovascular Risk Factors (DM, HTN, Dyslipidemia, smoking, family history of cardiovascular disease), Atrial fibrillation risk factors (CHADS-2 score; CHF, Age >75, DM, prior stroke/CVA), Prior atrial fibrillation ablation procedures, echocardiographic parameters (LVEF, Left atrial size), MRI parameters (Left ventricular end-diastolic volume, left ventricular end systolic volume, left ventricular stroke volume, LVEF, left atrial volume, right ventricular volumes and ejection fraction.)
qualitatively comparison with a standard scale | up to 6 weeks
  qualitatively comparison will be done for ECG signal quality and artifact between the 12-lead and 3-lead ECG arms using a standard scale. A 5 point Likert scale will be used with the below scores:
  1. indicating 12-lead ecg quality is substantially worse than 3-lead ecg
  2. somewhat worse
  3. equivalent
  4. somewhat better
  5. significantly better

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No